CLINICAL TRIAL: NCT06599398
Title: Bridging Hospital to Home for Children with Medical Complexity and Their Families: the Effectiveness of a Transitional Care Unit (the "Jeroen Pit Huis")
Brief Title: Bridging Hospital to Home for Children with Medical Complexity and Their Families
Acronym: BRIDGE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Erasmus Medical Center (Other); Stichting Katholieke Universiteit- Radboudumc (RUMC), Netherlands (Unknown); University Medical Center Groningen (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Clara van Karnebeek, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: BRIDGE
Record Dates: First submitted 2023-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Children with Medical Complexity
Keywords: Children with Medical Complexity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention group: The intervention group comprise patients and families who had an intermediate stay between hospital and home in the Jeroen Pit Huis (JPH)
  Interventions: Other: Jeroen Pit Huis
- Control groups: The control groups comprise patients and families who undergo the hospital to home transition directly from the hospital. This includes patients from the EMC, RUMC, and UMCG. Patients from the AUMC who transition directly from hospital to home without an intermediate stay in the JPH will also be included in the control group.
  Interventions: Other: Jeroen Pit Huis

INTERVENTIONS:
Other: Jeroen Pit Huis — The JPH is a unique and innovative Transitional Care Unit (TCU) situated in close proximity of the AUMC. In this TCU, patients and their family reside in separate private home-like apartments. The families can stay while practising in, and adapting to, their new reality until they are ready to transition home. A multidisciplinary team of healthcare experts (nurses, psychosocial care workers, family counsellors, and paediatricians) are gradually guiding parents towards taking on the role of their child's primary caregiver. This process is guided by a newly developed seven phase care path.One condition for staying in the JPH is that one parent is always present. In this form (24/7 parental stay and nursing care directly available under the supervision of pediatricians) the JPH is unique in the Netherlands.

SUMMARY:
The goal of this observational study is to evaluate an innovative pediatric transitional care unit called the Jeroen Pit Huis (JPH). The primary objective of our study is to investigate whether an intermediate stay between hospital and home in the JPH have a favourable effect on healthcare consumption, patient, parent and family-relevant quantitative outcome measures, compared to discharge directly from a hospital ward. Parents will be asked to complete several questionnaires on three different time points (at discharge, 3 and 12 months of follow up).

DETAILED DESCRIPTION:
Rationale: Children with Medical Complexities (CMC) often require 24/7 expert care for which often prolonged (re)admissions in a university medical centre (UMC) are necessary which, in turn, impedes discharge home. Hospital to home transitions of CMC is a multi-faceted process with many challenges and obstacles. This protocol describes the evaluation of an innovative Transitional Care Unit (TCU) called the Jeroen Pit Huis (JPH), that aims to supports this transition.

Hypothesis: We hypothesize that an intermediate stay between hospital and home in the JPH will have a favourable effect on healthcare consumption, patient, parent and family-relevant quantitative outcome measures, compared to discharge directly from a hospital ward.

Objective: The primary objective of our study is to investigate whether an intermediate stay between hospital and home in the JPH lowers parental distress compared to discharge directly from a hospital ward. Furthermore, the effect on quality of life (QoL) in children and parents, growth, family functioning, impact on parental employment, parental self-efficacy, anxiety, depression, sleep disturbance, posttraumatic stress (PTSD), care satisfaction, and healthcare consumption will be assessed with and without an intermediate stay in the JPH.

Study design: Multicenter quasi-experimental prospective cohort study

Study population: Patients (term newborns up to the age of 18 years) who; (1) are admitted in the hospital with (a deterioration of) a chronic complex condition (CCC) and/or have (expected) continuous dependence on technology after discharge; (2) require specialized medical and/or allied health care after discharge; (3) are medically stable and/or have a set treatment regime and; (4) are not yet ready to be discharged home due organization-, care- or family circumstances.

Intervention (if applicable): Not applicable, since the JPH is the standard of transitional care in the Amsterdam UMC.

Main study parameters/endpoints:

Primary outcome measure at TCU/hospital discharge, 3 and 12 months of follow-up

1. Parental distress

   Secondary outcome measures
2. Quality of Life of children at JPH/hospital discharge, 3 and 12 months of follow-up.
3. Growth parameters (weight, length, head circumference) at study inclusion, JPH/hospital discharge, 3 and 12 months of follow-up.
4. Impact of having a CMC on parents' Quality of Life and family functioning at JPH/hospital discharge, 3 and 12 months of follow-up
5. Impact on parental employment at 12 months of follow-up
6. Parental self-efficacy, anxiety, depression, sleep disturbance at JPH/hospital discharge, 3 and 12 months of follow-up.
7. Parental Posttraumatic Stress Disorder (PTSD) at 3 and 12 months of follow-up
8. Satisfaction of the parents with the received care at JPH/hospital discharge
9. Healthcare consumption during 12 months of follow-up

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects do not benefit personally from study participation. This non-therapeutic research with minors will have negligible risks. The main burden of participation in this study is the need to complete several questionnaires in total on three different time points. The expected required time-investment of the children and their caregivers is approximately 2.5 hours in total (around 50 minutes at 3 different time points). Furthermore, it requires time and effort from physicians to screen and patients for inclusion.

ELIGIBILITY:
Subject eligibility (or inclusion) criteria for this are as follows:

1. Age: at term (older than 37 weeks corrected gestational age) and younger than 18 years
2. Admitted to the hospital with (a deterioration of) a chronic complex condition (CCC) [30] and/or (expected) continuous dependence on technology after discharge (see ad 2 below).
3. Expected need of specialized medical and/or allied health care after discharge
4. A stable medical condition and/or a set treatment regimen (see below ad 4)
5. Discharge home not yet possible due to organization-, care- or family circumstances (see below ad 5)
6. Have given informed consent (consenting process is described in chapter 11.2 recruitment and consent)

Ad 2 chronic complex condition Fulfils criteria of a chronic complex condition (CCC) [30] and/or (expected) continuous dependence on technology after discharge.

A complex chronic condition (CCC) is defined according to Feudtner et al. (1) as "any medical condition that can be reasonably expected to last at least 12 months (unless death intervenes) and to involve either several different organ systems or one organ system severely enough to require specialty pediatric care and probably some period of hospitalization in a tertiary care center." Verlaat et al., updated the CCC list based on expert opinion [31]. A table of diagnosis classified as CCC can be found in appendix 1. An unknown but suspected complex and chronic condition, such as a child born with multiple congenital anomalies but lacking a unifying diagnosis, will be included.

Ad 4 stable medical condition

The patient is defined as being in a stable medical condition if there is:

1. A patent, safe airway to remain in the home situation, whether or not by means of a trachea cannula
2. Adequate respiration, whether or not by means of (intermittent) support with oxygen, non-invasive ventilation or invasive ventilation via a trachea cannula
3. A neurologically stable condition that may include temporary neurological impairments (such as seizures) not interfering (potentially life-threatening) with other vital functions such as respiration or circulation
4. Drug treatment that can be given at home where (if applicable): a nasogastric, duodenal or jejunal tube and/or a percutaneous endoscopic gastrostomy (PEG) tube is in situ, or if necessary, a 'home-proof' intravenous access is guaranteed
5. In case of enteral tube feeding, the nasogastric, duodenal or jejunal tube and/or a percutaneous endoscopic gastrostomy (PEG) tube is in situ, and the feeding schedule may be built up, reduced or variable if there are no contraindications for this. In case of parenteral feeding, the parenteral nutrition home program must be organized according to the home situation.

Ad 5 organization-, care- or family circumstances include the lack of 1 or more of the following requirements for safe discharge home:

1. A sustainable care plan using the four 'Medische Kindzorg Systeem' domains (medical, safety, development and social) has been drawn up that includes all four domains such as among others (Medical Child care System that is used in The Netherlands to structure medical child care in the home situation):

   * care needs
   * clear coordination of tasks and responsibilities of parents and healthcare professionals (primary, secondary and tertiary care).
2. The necessary medical and nursing care support (such as a feeding pump, adequate home care).
3. Parents know who to contact with questions about the organization of care (e.g. financial issues, wheelchair, municipality)
4. Essential medical technology is available at home and can be used for care.
5. Reimbursement of care at home is adequately arranged.
6. The house is located and furnished in such a way that the child can stay in it safely (accessibility for emergency services, telephone contact with parents, technical facilities)

   Parents/informal carers are adequately trained to take care of the child in the home situation, that means that they:
7. Master care in all areas (medical, nursing, technical, psychosocial)
8. Obtain declaration of care competencies, in particular:

   * assessment for somatic deterioration
   * acting in emergency situations (e.g. seeking help, resuscitation and if applicable: cannula dislocation, PEG probe problems, docking of a seizure)
   * realizing when to call for help and whom to call for help
9. Can obtain adequate telephone assistance (working telephone, English/Dutch speaking)
10. Are psychologically and emotionally ready to deal with new home situation (according to care professionals)

A potential subject will be excluded from participation in this study if:

1. The patient is in need of end-of-life care
2. Existence of predominantly social/family issues without serious medical problems in the index child
3. Patient with behavioural/psychiatric problems necessitating other type of care
4. Patient requiring rehabilitation medical care
5. Patients who are not directly discharged home from the hospital (except for the JPH (e.g. via de Boeg, Villa Expert Care))
6. Contagious disease that requires strict isolation

Ages: 0 Minutes to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population exists of all children admitted to one of the four UMCs. The population will be predominantly CMC. CMC have one or more chronic conditions, functional limitations, high family identified needs, and a high use of healthcare resources [1]. Eligible participants fulfil all inclusion and no exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Parental distress | Baseline, 3 and 12 months of follow-up
  Distress Thermometer for Parents (DT-P)

SECONDARY OUTCOMES:
Quality of Life of children | Baseline, 3 and 12 months of follow-up
  Generieke Patient Reported Outcome Measures (GPROM) voor Kinderen
Growth weight parameters | Study inclusion, baseline, 3 and 12 months of follow-up
  Weight in kilograms
Growth length parameters | Study inclusion, baseline, 3 and 12 months of follow-up
  height in meters
Impact of having a CMC on parents' Quality of Life and family functioning | Baseline, 3 and 12 months of follow-up
  PedsQL FiM
Impact on parental employment | 12 months of follow-up
  Self-constructed questionnaire
Parental self-efficacy | Baseline, 3 and 12 months of follow-up
  Parental Measure of Self-Efficacy Managing a Child's Medications and Treatments
Parental anxiety | Baseline, 3 and 12 months of follow-up
  The PROMIS v1.0 - Anxiety 4a
Parental depression | Baseline, 3 and 12 months of follow-up
  PROMIS v1.0 - Depression 4a short-forms
Parental sleep disturbance | Baseline, 3 and 12 months of follow-up
  Short form 4a PROMIS Sleep Disturbance (SD)
Parental Posttraumatic Stress Disorder (PTSD) | 3 and 12 months of follow-up
  PCL-5
Satisfaction of the parents with the received care | Baseline
  MPOC-20
Healthcare consumption - Length of hospital stay | During 12 months of follow-up
  Length of hospital stay in days
Healthcare consumption - Number of (PICU) readmissions | During 12 months of follow-up
  Number of (PICU) readmissions
Healthcare consumption - Emergency department visits | During 12 months of follow-up
  Emergency department visits
Healthcare consumption - (un)planned outpatient visits | During 12 months of follow-up
  (un)planned outpatient visits

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haspels HN, Mikkers MC, Knoester H, Jansen NJG, Ahout IML, Maaskant JM, van de Riet L, Haverman L, Dulfer K, Haasnoot M, Alsem MW, de Hoog M, van Woensel JBM, Joosten KFM, van Karnebeek CD; Transitional Care Unit Consortium. Bridging hospital to home for children with medical complexity and their families: an observational prospective cohort study protocol to assess the effectiveness of an innovative transitional care unit in the Netherlands (BRIDGE study). BMJ Open. 2025 Apr 19;15(4):e093693. doi: 10.1136/bmjopen-2024-093693. PMID 40254310